CLINICAL TRIAL: NCT04945642
Title: Phase 2 Study of High Dose-Rate Brachytherapy and Stereotactic Body Radiotherapy for Intermediate and High Risk Localized Prostate Adenocarcinoma (HYDRA)
Brief Title: High Dose-Rate Brachytherapy and Stereotactic Body Radiotherapy for the Treatment of Prostate Adenocarcinoma
Acronym: HYDRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-000704; NCI-2021-05623 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-14; First posted 2021-06-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Prostate Adenocarcinoma; Stage IIB Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (HDR-BT, SBRT) (Experimental): Patients undergo HDR-BT for up to 24 hours and undergo SBRT every other day or consecutive days for up to 14 consecutive chronologic days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: High-Dose Rate Brachytherapy; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: High-Dose Rate Brachytherapy — Undergo HDR-BT
  Other Names: Brachytherapy, High Dose
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial investigates the effect of high dose-rate brachytherapy and stereotactic body radiotherapy in treating patients with prostate adenocarcinoma. Brachytherapy, also known as internal radiation therapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the biochemical progression-free survival (b-PFS) at the 5-year time point after combination therapy of stereotactic body radiotherapy (SBRT) and high dose rate (HDR)-brachytherapy (BT) boost stratified by patients with intermediate and high-risk prostate cancer.

II. To estimate the rate of acute >= grade 3 patient-reported genitourinary (GU) and gastrointestinal (GI) symptoms determined within 90 days after treatment completion, respectively.

SECONDARY OBJECTIVES:

I. To estimate patient-reported GU symptoms at the end of radiotherapy and within 6, 12, 24, and 60 months from radiotherapy completion.

II. To estimate patient reported GI symptoms at the end of radiotherapy and within 6, 12, 24, and 60 months from radiotherapy completion.

III. To estimate the cumulative incidence of acute grade >= 2 GU physician-scored toxicity, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale.

IV. To estimate the cumulative incidence of acute grade >= 2 GI physician-scored toxicity, as assessed by the CTCAE version 5.0 scale.

V. To estimate the cumulative incidence of late >= 2 GU physician-scored toxicity, as assessed by the CTCAE version 5.0 scale.

VI. To estimate the cumulative incidence of late >= 2 GI physician-scored toxicity, as assessed by the CTCAE version 5.0 scale.

VII. To determine the prostate specific antigen (PSA) complete response rate (PSA nadir =< 0.3ng/mL) at 3 months following treatment of combination SBRT and HDR-BT boost regardless of testosterone recovery.

VIII. To determine clinical progression-free survival at 5-years. IX. To determine distant metastasis-free survival at 5-years. X. To determine overall survival at 5-years.

OUTLINE:

Patients undergo HDR-BT for up to 24 hours and undergo SBRT every other day or consecutive days for up to 14 consecutive chronologic days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 90 days, every 3 months for 24 months, and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand a written informed consent document, and the willingness to sign it
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* History/physical examination with digital rectal examination of the prostate within 8 weeks prior to registration
* Histologically confirmed intermediate- to high-risk prostate adenocarcinoma (T1c-T3b, PSA > 10, and/or Gleason score >= 7
* No evidence of disease beyond the prostate and/or seminal vesicles (i.e., no suspicious pelvic lymph nodes or presence of metastatic disease outside the pelvis)
* Prostate size =< 60cc
* International Prognostic Scoring System (IPSS) score =< 15
* Able to safely receive moderate sedation or general anesthesia

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years
* Regional lymph node involvement
* Evidence of distant metastases
* Previous radical surgery (prostatectomy) or cryosurgery or high-intensity focused ultrasound for prostate cancer
* Previous pelvic irradiation or prostate brachytherapy
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Patients with history of inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis), high predisposition for radio-toxicity compared to general population (i.e., ataxia telangiectasia), or at risk for major bowel surgery
* Transurethral resection of the prostate (TURP) procedure within 6 months of radiation treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical failure | Up to 5 years
  Will be based on Phoenix criteria (either a rise of 2 ng/mL or more above nadir prostate specific antigen [PSA], or patients not meeting this criterion but underwent salvage therapies). The biochemical progression free survival (b-PFS) will be defined from the date of completing radiotherapy to the date biochemical failure, death, or last follow-up, stratified by prostate cancer risk classification. Kaplan-Meier method will be used.
Patient-reported genitourinary (GU) and gastrointestinal (GI) symptoms | At 90 days
  Will be assessed on the Expanded Prostate Cancer Index-26 (EPIC-26) questionnaire.

SECONDARY OUTCOMES:
Patient-reported GU symptoms | At end of radiotherapy, 6, 12, 24, and 60 months
  Will be assessed on EPIC-26. EPIC assesses the disease-specific aspects of prostate cancer and its therapies within the genitourinary summary domain. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.
Patient-reported GI symptoms | At end of radiotherapy, 6, 12, 24, and 60 months
  Will be assessed on EPIC-26. EPIC assesses the disease-specific aspects of prostate cancer and its therapies within the gastrointestinal summary domain. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.
The acute grade >= 2 GU physician-scored toxicity | Up to 90 days from treatment completion
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The acute grade >= 2 GI physician-scored toxicity | Up to 90 days from treatment completion
  Will be assessed by CTCAE version 5.0.
The late grade >= 2 GU physician-scored toxicity | 90 days from treatment completion, assessed up to 5 years
  Will be assessed by CTCAE version 5.0.
The late grade >= 2 GI physician-scored toxicity | 90 days from treatment completion, assessed up to 5 years
  Will be assessed by CTCAE version 5.0.
PSA complete response | 3 months after treatment completion
  Will be defined as PSA =< 0.3 ng/mL three months after treatment completion.
Clinical disease progression to any anatomical site | Up to 5 years
  Will be based on patient history, physical examination, or imaging (computed tomography [CT], magnetic resonance imaging [MRI], positron emission tomography [PET]).
Clinical distant disease progression to anatomical sites outside prostate and regional lymph nodes | Up to 5 years
  Will be based on imaging (CT, PET).
Number of participants lost-to-follow-up | Up to 5 years
  Number of deaths or patients lost-to follow-up during the follow-up period
Progression-free survival | Up to 5 years
  Will be estimated by the Kaplan-Meier method.
Distant disease-free survival | Up to 5 years
  Will be estimated by the Kaplan-Meier method.
Overall survival | Up to 5 years
  Will be estimated by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Yoon, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California at Los Angeles / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States